CLINICAL TRIAL: NCT07241897
Title: DPP4 Inhibitor on Post-stroke Cognitive Impairment in Ischemic Stroke Patients With Type 2 Diabetes Mellitus (DISC-DM): Multicentre, Double Blind, Randomised, Placebo Controlled Trial
Brief Title: DPP4 Inhibitor Intervention on Post-stroke Cognitive Impairment in Ischemic Stroke Patients With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, yifang zhu, Professor, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LC2024019; 82471226 (Other Grant/Funding Number: the National Natural Science Foundation of China)
Record Dates: First submitted 2025-09-20; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke; Diabete Mellitus
Keywords: DPP4 inhibitors; Ischemic Stroke; PSCI; Diabetes Mellitus; RCT
MeSH Terms: conditions — Ischemic Stroke; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Intervention Group: Sentagliptin Phosphate 50 mg, once daily, plus metformin hydrochloride extended-release tablets (50 mg, two or three times daily). If blood glucose is still not well-controlled, sulfonylurea drugs may be added as needed.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Centralized network-based randomization will be used, with matching based on study center, patient age, gender, and glycated hemoglobin levels at the time of randomization. A double-blind design will be implemented, with patients randomly assigned in a 1:1 ratio to either the DPP4 inhibitor intervention group or the placebo control group, with both researchers and patients unaware of the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Sentagliptin Phosphate 50 mg, once daily, plus metformin hydrochloride extended-release tablets (50 mg, two or three times daily). If blood glucose is still not well-controlled, sulfonylurea drugs may be added as needed.
  Interventions: Drug: Sentagliptin Phosphate - single dose
- Control Group (Placebo Comparator): Placebo (identical in size, shape, color, appearance, and odor to Sentagliptin Phosphate, 50 mg, once daily) plus metformin hydrochloride extended-release tablets (50 mg, two or three times daily). If blood glucose is still not well-controlled, sulfonylurea drugs may be added as needed
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sentagliptin Phosphate - single dose — Sentagliptin Phosphate 50 mg, once daily, plus metformin hydrochloride extended-release tablets (50 mg, two or three times daily). If blood glucose is still not well-controlled, sulfonylurea drugs may be added as needed.
  Arms: Intervention Group
Drug: Placebo — Placebo (identical in size, shape, color, appearance, and odor to Sentagliptin Phosphate, 50 mg, once daily) plus metformin hydrochloride extended-release tablets (50 mg, two or three times daily). If blood glucose is still not well-controlled, sulfonylurea drugs may be added as needed.
  Arms: Control Group

SUMMARY:
Post-stroke cognitive impairment (PSCI) increases the risk of disability and mortality in stroke patients, thereby exacerbating the disease burden of stroke. Type 2 diabetes is a major risk factor for PSCI, and stroke patients with type 2 diabetes have a higher risk of developing PSCI. Despite the high incidence and severe impact of PSCI, effective intervention methods are still lacking. Identifying safe and effective drugs to improve cognitive function in stroke patients and reduce the risk of PSCI, especially for those with type 2 diabetes, is of significant importance and could help reduce the burden of stroke.

Dipeptidyl peptidase-4 (DPP4) inhibitors are first-line antidiabetic drugs, and several studies have shown that DPP4 inhibitors provide benefits beyond glucose control, including significantly improving cognitive function in patients with type 2 diabetes or slowing the progression of cognitive impairment. Our previous research found a significant negative correlation between baseline plasma soluble DPP4 (sDPP4) levels and the 90-day PSCI risk in ischemic stroke patients. Moreover, some studies indicate that DPP4 inhibitors can increase plasma sDPP4 levels. Based on this, we hypothesize that DPP4 inhibitors could be effective for PSCI intervention and may improve cognitive function post-stroke.

This project aims to conduct a multicenter, randomized, double-blind, placebo-controlled study. We will include patients with mild ischemic stroke combined with type 2 diabetes and provide continuous intervention with DPP4 inhibitors or a placebo for 180 days. Cognitive function in both groups will be assessed before and after intervention to determine if DPP4 inhibitors can improve cognitive function and reduce the risk of PSCI in ischemic stroke patients with type 2 diabetes. Clinical blood samples and imaging data will also be used to preliminarily explore potential mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Mild ischemic stroke, defined as a National Institutes of Health Stroke Scale (NIHSS) score ≤ 5.
2. Coexisting type 2 diabetes with a disease duration of less than 5 years.
3. Ability to complete the MoCA, MMSE, and the NINDS-CSN-recommended 1-hour standardized neuropsychological test for VCI.
4. Age between 40 and 75 years.
5. Onset of stroke within the last 2 weeks.
6. Glycated hemoglobin (HbA1c) between 6.5% and 8.5%.
7. More than 9 years of education.
8. Informed consent signed by the patient or their family.

Exclusion Criteria:

1. Coexisting dementia or severe cognitive impairment (MoCA < 17).
2. Coexisting severe depression, defined as a Hamilton Depression Rating Scale (HAMD) score ≥ 20.
3. Prior use of cognitive-enhancing drugs, such as donepezil or memantine.
4. Allergy to DPP4 inhibitors.
5. Past or current use of DPP4 inhibitors.
6. Past or current use of GLP-1 agonists.
7. Type 1 diabetes, latent autoimmune diabetes in adults, secondary diabetes, malignant tumors, autoimmune diseases, or other endocrine-related diseases.
8. Moderate or severe liver or kidney dysfunction.
9. Chronic or acute pancreatitis.
10. Pregnancy or lactation.
11. Severe infection or severely impaired immune response.
12. Participation in other clinical trials.
13. Past or current use of insulin therapy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in MoCA score before and after the 180-day intervention | 180 days
  Change in MoCA score before and after the 180-day intervention

SECONDARY OUTCOMES:
PSCI incidence at 180 days | 180 days
  MoCA score < 25
Changes in MMSE score and scores in various cognitive domains before and after the 180-day intervention | 180 days
  Changes in MMSE score and scores in various cognitive domains before and after the 180-day intervention
Changes in MoCA and MMSE scores before and after the 90-day intervention | 90 days
  Changes in MoCA and MMSE scores before and after the 90-day intervention
Modified Rankin Scale (mRS) score and cardiovascular and cerebrovascular events at 90 and 180 days | 90 days and 180 days
  Modified Rankin Scale (mRS) score and cardiovascular and cerebrovascular events at 90 and 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] You S, Bi Y, Miao M, Bao A, Du J, Xu T, Liu CF, Zhang Y, He J, Cao Y, Zhong C. Plasma sDPP4 (Soluble Dipeptidyl Peptidase-4) and Cognitive Impairment After Noncardioembolic Acute Ischemic Stroke. Stroke. 2023 Jan;54(1):113-121. doi: 10.1161/STROKEAHA.122.040798. Epub 2022 Dec 7. PMID 36475470
- [Result] You S, Miao M, Lu Z, Bao A, Du J, Che B, Xu T, Zhong C, Cao Y, Liu CF, Zhang Y, He J. Plasma Soluble Dipeptidyl Peptidase-4 and Risk of Major Cardiovascular Events After Ischemic Stroke: Secondary Analysis of China Antihypertensive Trial in Acute Ischemic Stroke (CATIS). Neurology. 2022 Aug 30;99(9):e925-e934. doi: 10.1212/WNL.0000000000200784. Epub 2022 Jun 2. PMID 35654589
- [Result] Baggio LL, Varin EM, Koehler JA, Cao X, Lokhnygina Y, Stevens SR, Holman RR, Drucker DJ. Plasma levels of DPP4 activity and sDPP4 are dissociated from inflammation in mice and humans. Nat Commun. 2020 Jul 28;11(1):3766. doi: 10.1038/s41467-020-17556-z. PMID 32724076
- [Result] Ma M, Hasegawa Y, Koibuchi N, Toyama K, Uekawa K, Nakagawa T, Lin B, Kim-Mitsuyama S. DPP-4 inhibition with linagliptin ameliorates cognitive impairment and brain atrophy induced by transient cerebral ischemia in type 2 diabetic mice. Cardiovasc Diabetol. 2015 May 20;14:54. doi: 10.1186/s12933-015-0218-z. PMID 25986579
- [Result] Chiazza F, Tammen H, Pintana H, Lietzau G, Collino M, Nystrom T, Klein T, Darsalia V, Patrone C. The effect of DPP-4 inhibition to improve functional outcome after stroke is mediated by the SDF-1alpha/CXCR4 pathway. Cardiovasc Diabetol. 2018 May 19;17(1):60. doi: 10.1186/s12933-018-0702-3. PMID 29776406
- [Result] Borzi AM, Condorelli G, Biondi A, Basile F, Vicari ESD, Buscemi C, Luca S, Vacante M. Effects of vildagliptin, a DPP-4 inhibitor, in elderly diabetic patients with mild cognitive impairment. Arch Gerontol Geriatr. 2019 Sep-Oct;84:103896. doi: 10.1016/j.archger.2019.06.001. Epub 2019 Jun 3. PMID 31204117
- [Result] Jeong SH, Kim HR, Kim J, Kim H, Hong N, Jung JH, Baik K, Cho H, Lyoo CH, Ye BS, Sohn YH, Seong JK, Lee PH. Association of Dipeptidyl Peptidase-4 Inhibitor Use and Amyloid Burden in Patients With Diabetes and AD-Related Cognitive Impairment. Neurology. 2021 Sep 14;97(11):e1110-e1122. doi: 10.1212/WNL.0000000000012534. Epub 2021 Aug 11. PMID 34380754
- [Result] Sun C, Xiao Y, Li J, Ge B, Chen X, Liu H, Zheng T. Nonenzymatic function of DPP4 in diabetes-associated mitochondrial dysfunction and cognitive impairment. Alzheimers Dement. 2022 May;18(5):966-987. doi: 10.1002/alz.12437. Epub 2021 Aug 10. PMID 34374497
- [Result] Zhong J, Maiseyeu A, Davis SN, Rajagopalan S. DPP4 in cardiometabolic disease: recent insights from the laboratory and clinical trials of DPP4 inhibition. Circ Res. 2015 Apr 10;116(8):1491-504. doi: 10.1161/CIRCRESAHA.116.305665. PMID 25858071
- [Result] Mulvihill EE, Drucker DJ. Pharmacology, physiology, and mechanisms of action of dipeptidyl peptidase-4 inhibitors. Endocr Rev. 2014 Dec;35(6):992-1019. doi: 10.1210/er.2014-1035. Epub 2014 Sep 12. PMID 25216328
- [Result] Levine DA, Wadley VG, Langa KM, Unverzagt FW, Kabeto MU, Giordani B, Howard G, Howard VJ, Cushman M, Judd SE, Galecki AT. Risk Factors for Poststroke Cognitive Decline: The REGARDS Study (Reasons for Geographic and Racial Differences in Stroke). Stroke. 2018 Apr;49(4):987-994. doi: 10.1161/STROKEAHA.117.018529. Epub 2018 Mar 16. PMID 29581343
- [Result] Rost NS, Brodtmann A, Pase MP, van Veluw SJ, Biffi A, Duering M, Hinman JD, Dichgans M. Post-Stroke Cognitive Impairment and Dementia. Circ Res. 2022 Apr 15;130(8):1252-1271. doi: 10.1161/CIRCRESAHA.122.319951. Epub 2022 Apr 14. PMID 35420911

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT07241897/SAP_000.pdf